CLINICAL TRIAL: NCT04978233
Title: Use of the Opal Patient Portal Application for Daily Follow-up of People at Home With COVID-19: The Opal-COVID Feasibility Study
Brief Title: The Opal - COVID-19 Study
Status: Completed | Type: Observational
Sponsor: Dr. Bertrand Lebouche (Other)
Responsible Party: Sponsor-Investigator, Dr. Bertrand Lebouche, Bertrand Lebouché MD, PhD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 2021-6763
Record Dates: First submitted 2020-12-03; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
Keywords: COVID-19; self-isolation; mHealth; patient portals
MeSH Terms: conditions — COVID-19 | interventions — Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MUHC COVID-19 patients: COVID-19 infected patients, newly diagnosed at the RI-MUHC
  Interventions: Other: sociodemographic and health, daily self-assessment, and feasibility of using the Opal app for COVID

INTERVENTIONS:
Other: sociodemographic and health, daily self-assessment, and feasibility of using the Opal app for COVID — The intervention consists of having confirmed COVID-19 infected participants register for the Opal app and complete a daily questionnaire on symptoms related to their physical and mental health as well as on certain key vital signs (e.g., oxygen saturation, heart rate, temperature). A nurse will check the questionnaire results each day and determine the need for a teleconsultation with an infectious disease physician. Participants will be followed up for a minimum of 14 days, depending on their symptoms.

SUMMARY:
In collaboration with involved healthcare professionals and a patient advisory committee, this study tests the feasibility of using the Opal smartphone app to daily capture self-reported physical and psychological symptoms and vital signs among 50 people who are self-isolating at home with COVID-19. A healthcare team at Montreal's MUHC will remotely monitor their condition and offer advice and teleconsultations, as needed.

DETAILED DESCRIPTION:
In the context of the current pandemic, guidelines were issued by public health authorities to follow the progression of COVID-19 in the community, identify and treat affected people, and limit transmissions. About 90% of people with COVID-19 only exhibit mild symptoms and recover. However, a small percentage of people experience serious symptoms and require hospitalization for severe shortness of breath or low oxygen levels. The current public health protocol is to identify people with COVID-19 and isolate them from others at home to prevent the virus from spreading. Currently, there is no consensus on how to effectively follow-up and treat individuals with COVID-19 who are self-isolating at home. Research is urgently needed. This pilot study will assess the feasibility of one strategy for home-based COVID-19 follow-up . The Opal app for COVID is a mobile application that will allow the completion of a daily symptom and vital sign follow-up questionnaire that will be monitored by a healthcare team. Educational material will also be provided through the app. The study will especially assess the acceptability and usability of the smartphone app.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Fluent in English and/or French
* Confirmed positive for PCR+ SARS-CoV-2
* Willing and able to understand the requirements of study participation and provide oral informed consent
* Access to a smartphone, tablet or computer at home
* Access to an internet connection at home or data plan on their smartphone
* Comfortable with the idea of using a new smartphone application to complete daily questionnaires, access educational material, and communicate with the healthcare team, or having someone to assist them with technology
* Prescribed self-isolation at home
* Proof of identity (passport, RAMQ, driver's license)

Exclusion Criteria:

* Have received a negative laboratory test result for the infection with COVID-19
* Confirmed negative for PCR+ SARS-CoV-2 and hospitalized
* Has any reason, in the opinion of the investigator, which would make the candidate inappropriate for participation in an investigative study involving a smartphone application
* Enrollment in any study involving an investigational drug for COVID-19 disease during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 infected patients, newly diagnosed at the RI-MUHC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in the acceptability of the Opal app for COVID-19 | from day 1 to day 14
  the Acceptability of Intervention Measure
Change in the usability of the Opal app for COVID-19 | from day 1 to day 14
  the Health Information Technology Usability Evaluation Scale

SECONDARY OUTCOMES:
Contact with the healthcare team | from day 1 to day 14
  Rate of participant contact with the healthcare team
Change in symptoms | from day 1 to day 14
  Self-reported symptoms of COVID-19, collected daily
Patient satisfaction with scheduled teleconsultations | from day 1 to day 14
  the Short Questionnaire for Out-of-Hours Care
Change in vital signs temperature | from day 1 to day 14
  Celcius degrees, collected daily
Change in vital signs respiration rate | from day 1 to day 14
  breaths per minute, collected daily
Change in vital signs oxygen saturation | from day 1 to day 14
  SpO2 %, collected daily
Change in vital signs heart rate | from day 1 to day 14
  beats per minute, collected daily
Change in vital signs blood pressure | from day 1 to day 14
  Systiolic/diastiolic mmHg, collected daily

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lebouché, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irizarry T, DeVito Dabbs A, Curran CR. Patient Portals and Patient Engagement: A State of the Science Review. J Med Internet Res. 2015 Jun 23;17(6):e148. doi: 10.2196/jmir.4255. PMID 26104044
- [Background] Drew DA, Nguyen LH, Steves CJ, Menni C, Freydin M, Varsavsky T, Sudre CH, Cardoso MJ, Ourselin S, Wolf J, Spector TD, Chan AT; COPE Consortium. Rapid implementation of mobile technology for real-time epidemiology of COVID-19. Science. 2020 Jun 19;368(6497):1362-1367. doi: 10.1126/science.abc0473. Epub 2020 May 5. PMID 32371477
- [Background] Kildea J, Battista J, Cabral B, Hendren L, Herrera D, Hijal T, Joseph A. Design and Development of a Person-Centered Patient Portal Using Participatory Stakeholder Co-Design. J Med Internet Res. 2019 Feb 11;21(2):e11371. doi: 10.2196/11371. PMID 30741643
- [Background] Houlding E, Mate KKV, Engler K, Ortiz-Paredes D, Pomey MP, Cox J, Hijal T, Lebouche B. Barriers to Use of Remote Monitoring Technologies Used to Support Patients With COVID-19: Rapid Review. JMIR Mhealth Uhealth. 2021 Apr 20;9(4):e24743. doi: 10.2196/24743. PMID 33769943
- [Derived] Lessard D, Engler K, Ma Y, Rodriguez Cruz A, Vicente S; Opal-COVID-19 Patient Expert Committee; Kronfli N, Barkati S, Brouillette MJ, Cox J, Kildea J, Hijal T, Pomey MP, Bartlett SJ, Asselah J, Lebouche B. Remote Follow-up of Self-isolating Patients With COVID-19 Using a Patient Portal: Protocol for a Mixed Methods Pilot Study (Opal-COVID Study). JMIR Res Protoc. 2022 Aug 18;11(8):e35760. doi: 10.2196/35760. PMID 35820054